CLINICAL TRIAL: NCT06126107
Title: Gain and Loss Framed Text Messaging to Reduce Drinking Among Older Adults
Acronym: GLOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0653-Hunter
Record Dates: First submitted 2023-11-01; First posted 2023-11-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Consumption
Keywords: Mobile Health; Text messaging; Behavioral economics; older adults
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants will be urn randomized according to gender, age and intensity of drinking to the three conditions collected at screening. They will be assigned to one of 3 text-messaging programs.
Who Masked: Participant
Masking Description: Participants will be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Loss-framed Messaging (Active Comparator): Daily text messages on the consequences of hazardous drinking (e.g., "Think of all you have lost as a result of drinking too much. Make today a day that sets the stage for change.")
  Interventions: Behavioral: Brief Normative Feedback; Behavioral: Loss-framed Text-messaging
- Gain-framed Messaging (Active Comparator): Daily text messages on the benefits of reducing drinking to safe guidelines (e.g., "Think of all you can achieve if you can control your drinking. Make today a day that sets the stage for change.")
  Interventions: Behavioral: Brief Normative Feedback; Behavioral: Gain-framed Text-messaging
- Gain-framed and Loss-framed Messaging (Active Comparator): Daily text messages that alternate between loss-framed (e.g., "Think of all you have lost as a result of drinking too much. Make today a day that sets the stage for change.") and gain-framed messaging (e.g., "Think of all you can achieve if you can control your drinking. Make today a day that sets the stage for change.")
  Interventions: Behavioral: Brief Normative Feedback; Behavioral: Loss-framed Text-messaging; Behavioral: Gain-framed Text-messaging

INTERVENTIONS:
Behavioral: Brief Normative Feedback — Once a participant has completed the assessment of their drinking during the baseline battery, the participant will receive brief normative feedback about how their drinking compares to their peers.
Behavioral: Loss-framed Text-messaging — Daily text-messages on the consequence of hazardous drinking.
  Arms: Gain-framed and Loss-framed Messaging; Loss-framed Messaging
Behavioral: Gain-framed Text-messaging — Daily text messages on the benefits of reducing drinking to safe guidelines.
  Arms: Gain-framed Messaging; Gain-framed and Loss-framed Messaging

SUMMARY:
The goal of this study is to evaluate effectiveness of scalable, tailored text- messaging programs for alcohol use among older adults. This study focuses on gain and loss framing of behavior change goals (i.e., the positives of change and the negatives of remaining with the status quo), critical components of behavioral science and health behavioral interventions. Loss-framing is used to motivate individuals to avoid future problems by focusing on the consequences of no change in behavior, and gain-framing is used to facilitate progress by focusing on the benefits of change. The investigators will design and evaluate three text-messaging programs using a randomized controlled trial: (A) Loss-framed messaging (B) Gain-framed messaging; and (C) Combined (loss and gain) messaging among a sample of 150 older adults with hazardous drinking. Participants will be randomized to one of the three conditions, each of which will include 8 weeks of text-messaging. During the study participants will completed assessments online and via text messages to track drinking.

DETAILED DESCRIPTION:
There is an urgent call for efficient and effective assessment, prevention, and intervention among older adults (age 50 and older) to reduce health risk of hazardous drinking, encourage healthy aging, and reduce burden on healthcare systems. Brief, low-burden, low-cost, digital interventions among older adults can answer this call. Text-messaging health interventions are considered an effective, scalable way to deliver behavioral health interventions, and they have been used as evidence-based solutions in primary care settings among older adults for behaviors other than alcohol use to supplement traditional care. Contrary to stereotypes, older adults use mobile technology, seek online and mobile interventions, and often engage longer compared to younger populations. The primary objective of the proposed study is to evaluate effectiveness of scalable, tailored text- messaging programs for alcohol use among older adults. This study focuses on gain and loss framing of behavior change goals (i.e., the positives of change and the negatives of remaining with the status quo), critical components of behavioral science and health behavioral interventions. Loss-framing is used to motivate individuals to avoid future problems by focusing on the consequences of no change in behavior, and gain-framing is used to facilitate progress by focusing on the benefits of change. The investigators will design and evaluate three text-messaging programs using a randomized controlled trial: (A) Loss-framed messaging (B) Gain-framed messaging; and (C) Combined (loss and gain) messaging among a sample of 150 older adults with hazardous drinking. Participants will be randomized to one of the three conditions, each of which will last 8 weeks. Participants will undergo cross- sectional online assessments (baseline, week 4, week 8 and week 16), and they will also complete a mobile assessment (via text message) once per week to track drinking. The effects of condition on drinking behavior will be compared at weeks 4, 8 and 16. In addition, attrition from the study will be closely tracked. Finally, the investigators will explore how the effects condition are impacted by gender and age (via moderation analysis).

ELIGIBILITY:
Inclusion Criteria:

* Be fluent in and able to read English at the eighth grade level
* Between the ages 50 and 85
* Have an estimated average weekly consumption of greater than, for women and men 65 and older, 12, or for men 64 and younger, 15 standard drinks per week
* Be willing to reduce their drinking to non-hazardous levels
* Be willing to provide informed consent
* Own a mobile phone with SMS capability and have an active email address.
* Be willing to receive and respond to up to 120 text messages total per month, as well as four online, web- based surveys.

Exclusion Criteria:

* Demonstrate physiological dependence on alcohol, as evidenced by current or a history of serious physical withdrawal symptoms (e.g., measured by SAWS)
* Present with significant substance use (greater than weekly use) or a current substance use disorder (for any substance other than alcohol, nicotine, or caffeine, measured by self report on Form-90 based questions)
* Present with a serious psychiatric illness or suicide risk, as measured by previous inpatient treatment, medications for mood disorder or psychosis, recent suicidality, and the PHQ-9.
* Unable to understand research study procedures as evidenced by failing a short quiz at the end of reviewing the consent form.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Weekly sum of standard drinks | baseline, week 4, week 8, and week 16
  Measure 1 of drinking, average of weekly sum of standard drinks
Weekly sum of heavy drinking days | baseline, week 4, week 8, and week 16
  Measure 2 of drinking, average of weekly heavy drinking days

SECONDARY OUTCOMES:
Percent adherence to daily drinking assessment via text messages | once daily, starting at baseline, lasting for 8 weeks
  Responses to text messages (via text message) are considered "adherence" to the daily drinking assessment. This measure is akin to compliance.
Percent adherence to weekly drinking assessment via web | once weekly, starting at baseline, lasting 8 weeks
  Responses to text messages (via text message) are considered "adherence" to the weekly drinking assessment. This measure is akin to compliance.
Percent willingness to continue the program for another 8 weeks | At week 8 assessment
  Participants are asked, "would you like to continue to receive text messages for the next 8 weeks?" If participants report yes, that is willingness to continue in the program. If no, then participants are not willing to continue in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Kuerbis, LCSW, PhD, Principal Investigator — Silberman School of Social Work at Hunter College City, University of New York
Locations (1):
- Hunter College of CUNY, New York, New York, United States